CLINICAL TRIAL: NCT05980026
Title: Omega-3 Fatty Acids Supplementation Improves Early-stage Diabetic Nephropathy and Subclinical Atherosclerosis in Pediatric Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nancy Samir Elbarbary, Prof. of Pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ain shams Pediatrics 202021
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral omega-3 fatty acids supplementation (Active Comparator): Intervention group included pediatric patients with diabetic nephropathy receiving oral omega-3 fatty acids supplementation on a daily basis.
  Interventions: Drug: oral omega-3 fatty acids supplementation
- Placebo comparator (Placebo Comparator): Placebo group or control patients received placebo that were similar in appearance to omega 3 fatty acids and the administered dose was as the same schedule as omega 3 fatty acids.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: oral omega-3 fatty acids supplementation — oral omega-3 fatty acids supplementation
  Arms: oral omega-3 fatty acids supplementation
Dietary Supplement: Placebo — Patients in placebo group received placebo that were similar in appearance to omega 3 fatty acids and the administered dose was as the same schedule as omega 3 fatty acids.
  Arms: Placebo comparator

SUMMARY:
The investigators conducted this randomized-controlled trial to assess the effect of oral omega-3 supplementation on glycemic control, lipid profile, albuminuria level, kidney injury molecule-1 (KIM-1) and carotid intima media thickness (CIMT) to participants who were pediatric patients with T1DM and diabetic nephropathy.

DETAILED DESCRIPTION:
Management of diabetic kidney disease (DKD) mainly consists of correction of hyperglycemia, hypertension and dyslipidemia as well as modification of lifestyle. Primary prevention represents prevention from normoalbuminuria to microalbuminuria, while secondary prevention represents prevention from microalbuminuria to macroalbuminuria. Multiple interventional managements with control of blood glucose, blood pressure and lipid, and smoking cessation can significantly improve the prognosis of cardiovascular events and slow down the progression of renal disease.

Omega-3 fatty acids are polyunsaturated fatty acids (PUFAs) derived from fish oil. Numerous studies have evaluated the potential beneficial effects of omega-3 fatty acids on inflammatory, autoimmune, and renal diseases. Due to their anti-inflammatory effects, omega-3 fatty acids have been suggested to protect against kidney damage. Omega-3 fatty acids can reduce proteinuria in patients with chronic glomerular disease and slow immunoglobulin A (IgA) nephropathy. However, the information about the effects of omega-3 fatty acids on kidney function, particularly in diabetic kidney disease still lacks consensus .

No previous study assessed the role of omega-3 fatty acids in diabetes associated complications in particular diabetic nephropathy and subclinical atherosclerosis among pediatric patients with T1DM and there is insufficient evidence to recommend its supplementation for those patients. Therefore, the investigators conducted this study to investigate the role of omega-3 fatty acids as an adjuvant therapy for participants who had diabetic nephropathy in children and adolescents with T1DM and assess its relation glycemic control, microalbuminuria, kidney injury molecule-1, lipid levels and carotid intima media thickness as an index for subclinical atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* patients with T1DM on regular insulin therapy.
* age from 12 to 18 years.
* disease duration at least 5 years.
* having diabetic nephropathy in the form of microalbuminuria (urinary albumin excretion [UAE] 30-299 mg/g creatinine).
* hemoglobin A1c (HbA1c) ≤8.5% (69 mmol/mol).
* persistent microalbuminuria was confirmed by abnormal two or three urine samples over a 3- to 6-months period prior to the study despite angiotensin converting enzyme inhibitors (ACE-Is)

Exclusion Criteria:

* patients with any clinical evidence of infection.
* patients with renal impairment due to causes other than diabetes.
* other diabetic complications than nephropathy.
* elevated liver enzymes.
* hyper- or hypo-thyroidism.
* intake of any vitamins or food supplements one month before study.
* participation in a previous investigational drug study within the three months preceding screening.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2023-01-14 (Actual)

PRIMARY OUTCOMES:
change in UACR (mg/g creatinine) level | 6 months
  Urinary albumin excretion rate(mg/g creatinine)

SECONDARY OUTCOMES:
change in KIM-1 level (ng/mL) | 6 months
  KIM-1 level((ng/mL)
change in HbA1c(%) | 6 months
  HbA1c%

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy Elbarbary, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The data will be available on request

REFERENCES:
- [Derived] Elbarbary NS, Ismail EAR, Mohamed SA. Omega-3 fatty acids supplementation improves early-stage diabetic nephropathy and subclinical atherosclerosis in pediatric patients with type 1 diabetes: A randomized controlled trial. Clin Nutr. 2023 Dec;42(12):2372-2380. doi: 10.1016/j.clnu.2023.10.007. Epub 2023 Oct 13. PMID 37862823